CLINICAL TRIAL: NCT05599113
Title: Evaluation of the Clinical Efficacy of Extracorporeal Shock Wave Therapy in Temporomandibular Joint Patients Having Disc Displacement With Reduction
Brief Title: Can Extracorporeal Shock Wave Therapy Be Effective in Temporomandibular Joint Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29.01.2020/14
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Temporomandibular Joint Disc Displacement, With Reduction; Extracorporeal Shock Wave Therapy
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal Shock Wave Therapy (Experimental): Extracorporeal shock wave therapy (ESWT) is an expedient remedy that is used in various joint and muscle pain treatments, is non-invasive, is well tolerated by patients, and has few side effects.
  Interventions: Device: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — Extracorporeal shock wave therapy (ESWT) is an expedient remedy that is used in various joint and non-invasive muscle pain treatments

SUMMARY:
The aim of this study is to evaluate the clinical efficacy of Extracorporeal Shock Wave Therapy (ESWT) in patients with Temporomandibular Joint (TMJ) with Reduced Disc Displacement, by comparing it with standard treatment.

Scientific Basis and Validity of Medical Research: Temporomandibular Joint Disorders (TMR) are disorders that can cause pain in the head and neck region, limitation in mouth opening, and difficulties even in daily activities (eating, speaking, chewing, yawning, etc.). These disorders have various causes such as malocclusion, emotional stress, parafunctional habits, synovitis, capsulitis, osteoarthritis and intra-articular irregularities. Almost 25% of the world's population has TMJ intra-articular irregularities and these are usually treated with non-surgical methods. If these methods are not successful, surgical treatments are generally used. These non-surgical treatments include many physical therapy interventions such as occlusal splints, medical treatments, bite plates, ultrasound and subcutaneous electrical nerve stimulation, and low-level laser therapies. With these intraorally used occlusal splints, a balanced occlusal contact is achieved without applying any force to the mandible in the resting position. Occlusal splints are available in different designs and different construction materials. The stabilization splint, which is one of the most commonly used occlusal splints, and the modified Hawley splint are appliances produced from hard materials. However, some researchers have commented that soft spints produced from resilient materials may also be useful in the distribution of excessive force formed in parafunctional habits. While there are studies stating that hard splints provide more successful results than soft splints in the functional problems of the chewing system, there are also studies reporting that they have similar efficacy on muscle pain after short-term use.

Extracorporeal shock wave therapy (ESWT), another physical therapy modality, used in the treatment of various joint and muscle pains; it is an advantageous treatment modality that is non-invasive, well tolerated by patients and has few side effects. This modality is also used in diseases of the TMJ and masticatory muscles in various sources. The availability of different non-standard treatment regimens and the few studies on the short-term results of ESWT applications make the use of ESWT in the treatment of TMJ diseases still unclear and new studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with reduced disc displacement according to DC/TMD examination criteria
* 18-70 years old
* No systemic disease that may have effects on masticatory muscles or TMJ
* Individuals who do not have any tooth loss other than 3. molar teeth and accept the treatments to be done

Exclusion Criteria:

* Individuals with total or distal extension partial dentures
* Individuals who have previously received medical, pharmacological, or any form of treatment for TMD
* Individuals with recent facial or cervical trauma
* Individuals with the syndrome who have the potential to affect any component of the stomagnatic system
* Individuals with parafunctional habits such as clenching or grinding their teeth.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
VAS pain score | At baseline
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | 1 week
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
VAS pain score | 2 week
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10.
Painless Maximum Active Mouth Opening | At baseline
  Measurement with one exception (pain-free opening), every time the patients moves his/her mouth vertically or excursively, he or she is instructed to move it as far as possible in that direction in milimeter.
Painless Maximum Active Mouth Opening | 1 week
  Measurement with one exception (pain-free opening), every time the patients moves his/her mouth vertically or excursively, he or she is instructed to move it as far as possible in that direction in milimeter.
Painless Maximum Active Mouth Opening | 2 week
  Measurement with one exception (pain-free opening), every time the patients moves his/her mouth vertically or excursively, he or she is instructed to move it as far as possible in that direction in milimeter.
Passive Forced Mouth Opening | At baseline
  Measurement of movements for range of motion and for joint sounds are made with actively pushed on by the examiner in milimeter.
Passive Forced Mouth Opening | 1 week
  Measurement of movements for range of motion and for joint sounds are made with actively pushed on by the examiner in milimeter.
Passive Forced Mouth Opening | 2 week
  Measurement of movements for range of motion and for joint sounds are made with actively pushed on by the examiner in milimeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyza Ünalan Değirmenci, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alshihri A. Translational Applications of Extracorporeal Shock Waves in Dental Medicine: A Literature Review. Biomedicines. 2022 Apr 14;10(4):902. doi: 10.3390/biomedicines10040902. PMID 35453651
- [Result] Falkensammer F, Arnhart C, Krall C, Schaden W, Freudenthaler J, Bantleon HP. Impact of extracorporeal shock wave therapy (ESWT) on orthodontic tooth movement-a randomized clinical trial. Clin Oral Investig. 2014 Dec;18(9):2187-92. doi: 10.1007/s00784-014-1199-0. Epub 2014 Feb 19. PMID 24549763
- [Result] Pfaff JA, Boelck B, Bloch W, Nentwig GH. Growth Factors in Bone Marrow Blood of the Mandible With Application of Extracorporeal Shock Wave Therapy. Implant Dent. 2016 Oct;25(5):606-12. doi: 10.1097/ID.0000000000000452. PMID 27504532
- [Derived] Keskin Tunc S, Unalan Degirmenci B, Bilen M, Toprak ME, Kaplan S, Turan M. Can extracorporeal shock wave therapy be effective in temporomandibular joint disorder?: A pilot study. Medicine (Baltimore). 2024 Oct 25;103(43):e40052. doi: 10.1097/MD.0000000000040052. PMID 39470554